CLINICAL TRIAL: NCT06699472
Title: A Prospective, Randomized, Controlled Clinical Study on the Prevention of VDC/IE Chemotherapy Related Myelosuppression in Patients with Ewing's Sarcoma Using Trilaciclib
Brief Title: A Prospective, Randomized, Controlled Clinical Study on the Prevention of Chemotherapy Related Myelosuppression in Patients with Ewing's Sarcoma Using Trilaciclib
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhiguo Luo, MD, PhD, Deputy chief of medical oncology, chief physician，Fudan University Shanghai Cancer Center, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2409305-18
Record Dates: First submitted 2024-11-05; First posted 2024-11-21 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Ewing Sarcoma; Myelosuppression
Keywords: Ewing Sarcoma; Myelosuppression; CDK4/6 inhibitor; Chemotherapy
MeSH Terms: conditions — Sarcoma, Ewing | interventions — Drug Therapy; trilaciclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Chemotherapy+Trilaciclib (Experimental): Receive VDC+IE alternating chemotherapy combined with Trilaciclib, with 3 weeks as one course of treatment, for a total of 17 cycles or until disease progression and intolerable toxicity occur.
  Interventions: Drug: Chemotherapy; Drug: Trilaciclib Injection [Cosela]
- Chemotherapy (Active Comparator): Receive VDC+IE alternating chemotherapy with 3 weeks as one course of treatment, for a total of 17 cycles or until disease progression and intolerable toxicity occur.
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Drug: Chemotherapy — Vincristine (V), intravenous injection, 1.5 mg/m2 (maximum not exceeding 2mg), D1, odd cycle administration Doxorubicin (D), intravenous infusion, 75mg/m2, D1, odd cycle administration When the cumulative dose of doxorubicin is ≥ 375mg/m2, replace it with actinomycin D 1.25mg/m2 Cyclophosphamide (C), intravenous infusion, 1200mg/m2, D1, odd cycle administration Ifosfamide (I), intravenous infusion, 1800mg/m2, D1-5, even cycle administration Etoposide (E), intravenous infusion, 100mg/m2, D1-5, even cycle administration
  Other Names: VDC/IE alternating chemotherapy
Drug: Trilaciclib Injection [Cosela] — Trilaciclib, intravenous infusion, 240 mg/m2, administered following chemotherapy (2 hours after completion of vincristine administration and within 4 hours before administration of other chemotherapy drugs)
  Arms: Chemotherapy+Trilaciclib

SUMMARY:
This study is a prospective, open label, randomized controlled clinical trial aimed at patients with Ewing's sarcoma who have not received systematic anti-tumor treatment in the past. The aim is to evaluate the efficacy and safety of prophylactic use of Trilaciclib before VDC+IE chemotherapy.

Patients with Ewing's sarcoma who have not received systemic anti-tumor therapy in the past will be screened for qualified subjects who meet the inclusion criteria after signing informed consent. Eligible patients will be randomly divided into an experimental group and a control group in a 1:1 ratio. The control group will receive alternating VDC+IE chemotherapy for 3 weeks, a total of 17 cycles, or until disease progression, intolerable adverse reactions, or withdrawal of informed consent occur. The experimental group received VDC+IE alternating chemotherapy combined with Trilaciclib, with 3 weeks as one course of treatment, for a total of 17 cycles or until disease progression, intolerable toxicity, withdrawal of informed consent, initiation of other anti-tumor treatments, death, or other situations specified in the protocol where treatment should be discontinued. Both the control group and the experimental group can receive supportive nursing treatment according to clinical needs.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 14 years old and ≤ 40 years old;
* Histologically confirmed Ewing's sarcoma;
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) score of 0 to 1;
* Have not received any anti-tumor treatment other than surgery in the past;
* Expected survival of more than 3 months;
* Possess sufficient organ and bone marrow function, with laboratory test values meeting the following requirements within 7 days prior to enrollment (no blood components, cell growth factors, albumin, or other corrective treatment drugs are allowed within 14 days prior to obtaining laboratory tests), as follows Blood routine: Absolute neutrophil count (ANC) ≥ 1.5 × 109/L, platelet count (PLT) ≥ 100 × 109/L, hemoglobin (HGB) ≥ 100 g/L (no transfusion or erythropoietin dependence within 14 days) Liver function: serum total bilirubin ≤ 1.25 times the upper limit of normal (ULN); ALT and AST ≤ 2.5 x ULN (≤ 5x ULN for patients with liver metastases); Serum albumin ≥ 30 g/L; Alkaline phosphatase (ALP) ≤ 5 × ULN.

Renal function: Serum creatinine (Cr) ≤ 1.25 × ULN, or creatinine clearance rate ≥ 60 mL/min (using the standard Cockcroft Gault formula): Urine routine results show urinary protein<2+; For patients whose baseline urine routine test shows urinary protein ≥ 2+, 24-hour urine collection should be performed with a 24-hour urine protein quantification of<1g.

Coagulation function: International normalized ratio (INR) or prothrombin time (PT) ≤ 1.5 times ULN; If the subject is receiving anticoagulant therapy, as long as the INR is within the intended range of use of the anticoagulant drug.

* For female subjects of childbearing age, a urine or serum pregnancy test should be conducted 3 days before receiving the first study drug and the result should be negative;
* The subjects and their sexual partners are required to use a medically approved contraceptive measure (such as intrauterine device, contraceptive pill, or condom) during the study treatment period and within 6 months after the end of the study treatment period.

Exclusion Criteria:

* Previously received anti-tumor treatment other than surgery and radiation therapy for any malignant tumor;
* Subjects who cannot accept or tolerate this chemotherapy regimen for various reasons;
* Biopsy confirmed a patient with bone marrow infiltration;
* The patient has undergone significant surgical procedures unrelated to Ewing's sarcoma within the 4 weeks prior to enrollment, or has not fully recovered from such surgical procedures;
* Serious heart disease or discomfort, including but not limited to the following diseases:

Diagnosed history of heart failure or systolic dysfunction (LVEF<50%); High risk uncontrolled arrhythmias, such as atrial tachycardia, resting heart rate>100bpm, significant ventricular arrhythmias (such as ventricular tachycardia), or higher-level atrioventricular block (i.e. Mobitz II second or third degree atrioventricular block); Angina requiring treatment with anti angina drugs; Clinically significant heart valve disease; ECG shows transmural myocardial infarction; Poor control of hypertension (systolic blood pressure>180mmHg and/or diastolic blood pressure>100mmHg)

* Individuals with a known history of allergies to the components of this medication regimen;
* Breastfeeding female patients, female patients with fertility and positive baseline pregnancy test results, or reproductive age patients who are unwilling to take effective contraceptive measures during the entire trial period and within 7 months after the last study medication;
* The researchers believe that the patient is not suitable to participate in any other circumstances of this study.

Ages: 14 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 22 (Estimated)
Dates: Start 2024-10-31 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Duration of 4th degree neutropenia in the first treatment cycle | From enrollment to the end of Cycle 1 (each cycle is 21 days)

SECONDARY OUTCOMES:
The time for neutrophil count to recover to ≥ 0.5 × 10^9/L in the first treatment cycle | From enrollment to the end of Cycle 1 (each cycle is 21 days)
The incidence of febrile neutropenia during the first to fourth treatment cycles | From enrollment to the end of Cycle 4 (each cycle is 21 days)
The incidence of grade 3 or higher neutropenia in the first to fourth treatment cycles | From enrollment to the end of Cycle 4 (each cycle is 21 days)
The incidence of grade 3 or higher thrombocytopenia in the first to fourth treatment cycles | From enrollment to the end of Cycle 4 (each cycle is 21 days)
The incidence of grade 3 anemia or above during the first to fourth treatment cycles | From enrollment to the end of Cycle 4 (each cycle is 21 days)
The number of times and frequency of reduction of all cause chemotherapy drugs | From enrollment to the end of Cycle 4 (each cycle is 21 days)
The number of cycles of the first reduction of chemotherapy drugs | From enrollment to the end of Cycle 4 (each cycle is 21 days)
The incidence of infectious serious adverse events | From enrollment to the end of Cycle 4 (each cycle is 21 days)
EFS | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  Event Free Survival

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cencer Center,, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No